CLINICAL TRIAL: NCT01303666
Title: Tidal Irrigation Versus Intra-articular Steroid Injection in the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Dr Jo Ledingham, Portsmouth Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEO118
Record Dates: First submitted 2011-01-27; First posted 2011-02-25 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Craniospinal Irradiation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- TI of the knee (Active Comparator)
  Interventions: Procedure: TI of the knee
- Intra-articular CSI (Active Comparator)
  Interventions: Procedure: Intra-articular CSI

INTERVENTIONS:
Procedure: Intra-articular CSI — After full aseptic preparation, 40 mg triamcinolone acetonide and 2 ml 1% lignocaine were injected into the joint cavity using the medial patello-femoral approach via a 21-gauge needle.
  Arms: Intra-articular CSI
Procedure: TI of the knee — This was done as a day case procedure under local anaesthetic. The medial patello-femoral approach was used. After full aseptic preparation, the skin and soft tissues were infiltrated with 5e10 ml of 1% lignocaine. The joint was then instilled with a further 10 ml of 1% lignocaine.
  After an initial puncture using a scalpel, a 3.2 mm diameter wrist arthroscope was advanced into the joint cavity. Up to 1 l of 0.9% normal saline was then irrigated through the joint: saline was run into the joint until fully distended and then allowed to flow out of the joint in a cyclical method until the aspirated fluid runs clear for at least three successive cycles.
  Arms: TI of the knee

SUMMARY:
Previous studies have indicated that patient expectations, beliefs and preferences may have an impact on treatment outcomes. The KIVIS study was primarily designed to compare two effective treatments for knee osteoarthritis (tidal irrigation (medical washout of the knee) or intra-articular corticosteroid injection). At study entry any preference expressed by the patient for each of the treatment interventions was recorded. This study assessed the effects of two treatments given at a single time-point and hence the effects of patient preference could be assessed independently of any compliance issues.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of knee OA
* Knee pain for most days of the prior month
* Radiographic evidence consistent with knee OA
* Aged between 40 and 90 years old

Exclusion Criteria:

* Symptomatic hip OA
* Co-existent inflammatory or crystal arthritis
* Prior knee surgery
* Injury to the knee in the preceding 6 months
* Any intra-articular injection in the preceding 3 months
* Inability to provide informed consent

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2000-11; Primary Completion 2003-07 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
WOMAC pain (WP)score | Weeks 0
Visual Analogue Scale | Weeks 0
WOMAC pain (WP)score | Weeks 2
WOMAC pain (WP)score | Weeks 4
WOMAC pain (WP)score | Weeks 12
WOMAC pain (WP)score | Weeks 26
Visual Analogue Scale | Weeks 2
Visual Analogue Scale | Weeks 4
Visual Analogue Scale | Weeks 12
Visual Analogue Scale | Weeks 26

SECONDARY OUTCOMES:
WOMAC physical function score (WF) | Weeks 0,2,4,12,26
Overall assessment of the impact of the procedure by the patient (five point scale) (PA) | Weeks 0,2,4,12,26
Overall assessment of the impact of the procedure by the blinded clinician (five point scale)(CA) | Weeks 0,2,4,12,26
Time to walk fifty metre | Weeks 0,2,4,12,26
Analgesic intake | Weeks 0,2,4,12,26
Side effects of the procedure | Weeks 0,2,4,12,26

CONTACTS AND LOCATIONS:
Overall Officials: Nigel K Arden, Principal Investigator — MRC Epidemiology Resource Centre, Southampton General Hospital, Southampton, UK